CLINICAL TRIAL: NCT05671341
Title: Comparison of Balance, Activity-specific Balance Confidence and Quality of Life in Parkinson's Patients with Freezing and Relationship Between Neutrophil/lymphocyte Ratio
Brief Title: Comparison of Balance, Activity-specific Balance Confidence and Quality of Life in Parkinson's Patients
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Asli Demirtaş, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 2022/106
Record Dates: First submitted 2023-01-01; First posted 2023-01-04 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Balance; Balance confidence; Quality of life; Freezing; Neutrophil/Lymphocyte ratio
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parkinson's Patients with Motor Freezing: Individuals with Parkinson's Disease with motor freezing were included in this group.
  Interventions: Diagnostic Test: Assessment
- Parkinson's Patients Without Motor Freezing: Individuals with Parkinson's Disease without motor freeze were included in this group.
  Interventions: Diagnostic Test: Assessment

INTERVENTIONS:
Diagnostic Test: Assessment — Tandem walking test, Tandem Stance test, Activity-specific Balance Confidence Parkinson's Disease Quality of Life-8 N/L ratio Tinetti Balance Test UPDRS

SUMMARY:
Parkinson's disease is characterized by cardinal motor signs and motor freezing, gait, posture and balance disorder. About 80% of the causes of falls in Parkinson's patients are due to postural instability and motor freezing, and patients' quality of life is significantly affected. Loss of balance and falls, which are frequently experienced in Parkinson's patients, cause individuals to feel insecure during activities. It is thought that the quality of life of PD patients whose movements are restricted due to the fear of falling may also be negatively affected. The neutrophil/lymphocyte ratio is a marker of peripheral inflammation. The relationship of peripheral inflammation to balance, activity-specific balance confidence, and quality of life in individuals is unclear. The aim of this study was to compare balance, activity-specific balance confidence, quality of life, and the relationship between neutrophil/lymphocyte ratio in Parkinson's patients with and without freezing.

DETAILED DESCRIPTION:
Parkinson's disease is characterized by cardinal motor signs and motor freezing, gait, posture and balance disorder. About 80% of the causes of falls in Parkinson's patients are due to postural instability and motor freezing, and patients' quality of life is significantly affected. Loss of balance and falls, which are frequently experienced in Parkinson's patients, cause individuals to feel insecure during activities. It is thought that the quality of life of PD patients whose movements are restricted due to the fear of falling may also be negatively affected. The neutrophil/lymphocyte ratio is a marker of peripheral inflammation. The relationship of peripheral inflammation to balance, activity-specific balance confidence, and quality of life in individuals is unclear.

The aim of this study was to compare balance, activity-specific balance confidence, quality of life, and the relationship between neutrophil/lymphocyte ratio in Parkinson's patients with and without freezing.

A total of 20 Parkinson's Disease age of older the 50 participate in the research. Participants were divide into two groups with and without freezing.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with idiopathic Parkinson's disease
* Healthy individuals who do not have musculoskeletal disease or any neurological disease that may affect assessments
* Older than 50 years old
* Volunteer to participate in the study
* Grade 1-3 on the Modified Hoehn-Yahr Scale
* To have a score above 24 in the Standardized Mini Mental Test
* To have a hemogram follow-up in the last 1 month before the date of participation in the study.
* Being able to walk independently on flat ground

Exclusion Criteria:

* Having an additional or psychiatric disease other than Parkinson's disease
* Lack of cooperation
* Presence of orthopedic problems (such as fractures, osteoporosis, osteomyelitis)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients who applied to Nigde Omer Halisdemir University Training and Research Hospital Neurology Clinic will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Freezing of Gait Questionnaire | Baseline
  The scale is a scale that evaluates motor freezing in Parkinson's patients. It is questioned whether freezing occurs during activities such as walking and turning on the 6-item scale developed. In addition, in the presence of freezing, the severity, frequency and duration of freezing are recorded. The higher the score, the higher the freezing.
The Tinetti Balance and Gait Test | Baseline
  It provides useful information on the ability of sick individuals to comfortably perform various functional tasks. For this reason, it is an easily and inexpensively applicable scale. This test consists of two parts and a total of 16 questions. These are walking in the 7-question part and balance in the 9-question part. The total score in the first 9 questions constitutes the balance score, and the total score in the next 7 questions constitutes the walking score. The total score in balance and walking constitutes the TDYT total score. TDYT score calculation is done by observation. 2 points indicate that the movement is performed correctly, 1 point indicates that there are adaptations in the movement, and 0 points indicate that the desired movement cannot be performed. A total score of 18 or less after TDYT indicates a high fall risk, a score of 19-24 indicates a moderate fall risk, and a score above 24 indicates a low risk of falling.
Activity-Specific Balance Confidence | Baseline
  Individuals are asked 16 questions about daily living activities inside and outside the home. For each question, individuals are asked to rate their confidence in the activity between 0 and 100%. These values are added together and divided by 16 and the nearest decimal value is accepted as the value of the scale. The higher the score, the higher the balance confidence of individuals.
Parkinson's Disease Quality of Life-8 | Baseline
  One question from each of the eight domains in PHA-39, which are activities of daily living, physical discomfort, cognition, communication, emotional well-being, mobility, social support and stigma, gives the total domain score.Each question is scored between 0-4 points and points are added up. The total score is then divided by the total possible score and given as a percentage point out of 100. The lower the score, the higher the quality of life.
Hemogramme | Baseline
  The neutrophil/lymphocyte ratio is a marker of peripheral inflammation.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | Baseline
  This scale was created to evaluate the motor performance, mental and mental status, and activities of daily living of Parkinson's patients. It also evaluates motor fluctuations, dyskinesias, and autonomic dysfunction. The scale was prepared as 4 parts and 42 items. When the extremities are evaluated separately, it increases up to 55 items. Items are rated from 0 (no symptoms or signs) to 4 (most severe symptoms and signs). The first part evaluates the non-motor features of the disease, such as thoughts, behaviors, and emotions. The second part consists of activities of daily living. In the third part, motor examination, in the fourth part, the complications of the treatment are given. It is used to evaluate the symptoms of the disease and the complications that develop due to treatment. In this scale, which consists of 4 parts, the scoring of each item is between 0-4 points. The increase in the total score reflects the increase in the severity of the symptoms.
Tandem stance test: | Baseline
  During the tandem stance test, which allows the evaluation of static balance, the individual will be asked to position the heel of one of his feet to the tip of the other. While the individual maintains this position without support, the time elapsed until the individual's balance is broken will be recorded with the help of a stopwatch. For individuals without balance problems, the test takes 30 seconds. It will be continued until it is full.
Tandem walking test | Baseline
  The tandem walking test is a clinical assessment of dynamic balance associated with falls in many studies. It is recommended as a simple tool to identify those at risk of falling. The participant is asked to walk 10 steps in a straight line with the heel of one foot touching the toe of the other foot, with his hands folded over the chest, wearing comfortable shoes, and the time is recorded.

OTHER OUTCOMES:
Standardized Mini Mental Test | Baseline
  There are 19 items in this test, which consists of 5 main parts: orientation, recording memory, attention and calculation, recall and language. The total score of the test is evaluated out of 30 and 24 points are accepted as the threshold value for the diagnosis of mild dementia. The higher the score, the higher the cognition of individuals.
Modified Hoehn and Yahr Scale | Baseline
  This staging scale was developed by Margaret Hoehn and Melvin Yahr (1967) for use in describing the stage of Parkinson's disease. According to the staging scale, the disease is handled in 8 stages. The lower the stage, the better of the stage Parkinson's disease.
  Stage 0: No signs of disease Stage 1: Unilateral disease Stage 1.5: Unilateral plus axial involvement. Stage 2: Bilateral disease, no balance disorder. Stage 2.5: Mild bilateral disease recovering on pull test. Stage 3: Mild to moderate bilateral disease and some postural instability, physically independent.
  Stage 4: Severe disability, able to stand and walk unaided. Stage 5: Unassisted wheelchair or bed dependent.

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University Treaning and Research Hospital, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No